CLINICAL TRIAL: NCT03684915
Title: Clinical Post-operative Assessment of Chronic Signs & Symptoms Related to Infected Primary Molars After Using Rotary Versus Manual Systems in Cleaning the Root Canals: A Randomized Clinical Trial
Brief Title: Clinical Post-operative Assessment of Chronic Signs & Symptoms Related to Infected Primary Molars After Using Rotary Versus Manual Systems in Cleaning the Root Canals
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Basma Mohamed Zakaria Ahmed Zain, Principal investigator (Master Degree Student), Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-08-26
Record Dates: First submitted 2018-09-10; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Chronic Infection
Keywords: Rotary instrumentation; pulpectomy; primary teeth
MeSH Terms: conditions — Persistent Infection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rotary files (Experimental): 1. Pre-operative radiograph showing all roots and their apices.
  2. Local anaesthetic (to enable use of rubber dam clamp).
  3. Rubber dam isolation.
  4. Removal of caries.
  5. Removal of roof of pulp chamber.
  6. Removal of any remains of coronal pulp tissue with sharp sterile excavator or large bur in slow hand piece.
  7. Identify root canals.
  8. Irrigate with normal saline (0.9%)
  9. Estimate working lengths of root canals keeping 2 mm short of the radiographic apex.
  10. Insert rotary files into canals and debride the canals lightly and gently.
  11. Irrigate the root canals.
  12. Dry canals with pre-measured paper points, keeping 2 mm from root apices.
  13. Canals will be dried with paper points, obturated by injecting Metapex. (Meta Biomed - Metapex Root Canal Filling Material)
  14. Stainless steel crown will be performed
  Interventions: Device: Rotary files
- manual files (Active Comparator): All steps as that of intervention group are to be followed except step (j) instead of it; a manual files will be inserted into the canals for debridement lightly and gently
  Interventions: Device: Rotary files

INTERVENTIONS:
Device: Rotary files — using rotary files in cleaning root canals of infected primary molars

SUMMARY:
One of the most important concerns in pediatric dentistry is the loss of necrotic primary molars leading to space loss. pulpectomies for primary teeth with severe pulpal involvement should be considered as the treatment of choice.

Bacteria plays an essential role in the initiation and perpetuation of pulpal and periapical disease. The investigator's target when cleaning and shaping the root canal system is to remove bacteria-containing tissue.

The removal of organic debris is the main purpose of instrumentation in pulpectomy procedures in primary teeth, this could be achieved using manual or rotary Ni-Ti files. A practical pulpectomy technique for the primary teeth should include the following:1) Fast procedure with short treatment time and minimal number of appointments.2) Effective debridement of the root canal without weakening the tooth structure or endangering the underlining permanent teeth.3) Minimal procedural complications. 4) Maintaining tooth function until it is naturally exfoliated.

Manufacturers using rotary files highlight their cleaning efficiency for root canal preparations, simple procedures, and decreased procedure time, which is especially important in children.

Considering that preparation time is an important clinical factor in pediatric patient management, the use of rotary instruments for pulpectomies in primary teeth is recommended.

ELIGIBILITY:
Inclusion Criteria:

* primary molars with fistula / chronic abscess
* teeth which if lost possibility of space maintainer construction exists
* pre-operative radiograph showing absence of severe root resorption

Exclusion Criteria:

* teeth with non-restorable crowns
* expected shedding time within one year

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Resolution of fistula | 3 months
  unit of measurement: Yes/No using visual examination

SECONDARY OUTCOMES:
assessment of tooth mobility | 3 months
  unit of measurements : grades from 0-3 ,assessed by moving the tooth using two instruments ,one on the facial & the other on the lingual surfaces of the tooth

IPD SHARING:
Plan to Share IPD: Undecided